CLINICAL TRIAL: NCT06234995
Title: Cortical Electrophysiology of Response Inhibition in Parkinson's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Svjetlana Miocinovic, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00007291; P50NS123103 (NIH)
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Deep brain stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Intervention Model Description: Healthy controls and persons with PD will be compared in Aim 1. In Aim 3, participants with PD, who have had DBS leads implanted will complete study assessments under four different DBS stimulation settings.
Who Masked: Outcomes Assessor
Masking Description: A motor exam will be performed and video recorded for blinded analysis by a movement disorders neurologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Patients with Parkinson's Disease (Experimental): Patients with PD complete motor response inhibitions tasks under multiple conditions, depending on the study aim they are participating in. Those who are participants in Aim 1 of the study are able to also participate in Aims 2 and 3 if they are having a clinically indicated DBS leads implanted. Patients with PD will participate in the study for approximately 18 months which includes one preoperative visit, intraoperative data collection and two post-operative visits. As part of the motor inhibition tasks, EEG signals will be recorded. A cap similar to a swim cap will be placed on the head of the subject, and gel will be applied to the hair to get a good signal. Electrodes will be attached to the cap for recording of brain signals. A few additional flat electrodes will be placed on the skin to record hand muscle activity (for GNG task) and near the eyes to record eye movements. Accelerometer sensors will be utilized to record arm movements (for MSS task).
  Interventions: Drug: Levodopa; Device: Clinical DBS Setting; Device: Sham DBS; Device: DBS Setting Maximizing Prefrontal Activation; Device: DBS Setting Minimizing Prefrontal Activation
- Healthy Controls (No Intervention): Healthy participants complete motor response inhibition tasks during two study visits. Healthy controls will participate for approximately one month, which includes two study visits. As part of the motor inhibition tasks, EEG signals will be recorded. A cap similar to a swim cap will be placed on the head of the subject, and gel will be applied to the hair to get a good signal. Electrodes will be attached to the cap for recording of brain signals. A few additional flat electrodes will be placed on the skin to record hand muscle activity (for GNG task) and near the eyes to record eye movements. Accelerometer sensors will be utilized to record arm movements (for MSS task).

INTERVENTIONS:
Drug: Levodopa — Participants will take levodopa in dosages prescribed by their care provider. Patients will be instructed to not take their regularly prescribed PD medications for 12 hours prior to the study assessment, as is typical for clinical evaluations in patients with PD. Participants will be tested in both levodopa-off (after 12 hours of not having medication) and levodopa-on states.
  Other Names: L-Dopa
  Arms: Patients with Parkinson's Disease
Device: Clinical DBS Setting — Deep brain stimulation performed with the patients' optimized clinical setting.
  Arms: Patients with Parkinson's Disease
Device: Sham DBS — Deep brain stimulation performed with sham stimulation.
  Arms: Patients with Parkinson's Disease
Device: DBS Setting Maximizing Prefrontal Activation — Deep brain stimulation performed to maximize the activation of the prefrontal cortico-STN projections.
  Arms: Patients with Parkinson's Disease
Device: DBS Setting Minimizing Prefrontal Activation — Deep brain stimulation performed to minimize the activation of the prefrontal cortico-STN projections.
  Arms: Patients with Parkinson's Disease

SUMMARY:
Patients with Parkinson's Disease will be studied before, during, and after a deep brain stimulation implantation procedure to see if the stimulation location and the size of the electrical field produced by subthalamic nucleus (STN) DBS determine the degree to which DBS engages circuits that involve prefrontal cortex executive functions, and therefore have a direct impact on the patient's ability to inhibit actions.

DETAILED DESCRIPTION:
Patients with Parkinson's disease (PD) commonly develop difficulties with executive function due to neurodegeneration in neuronal networks that involve the prefrontal cortex and associative territories of the basal ganglia, even in early stages of the disease. Executive cognitive functions serve to direct behavior toward a goal and modify actions to accommodate changing demands. One of the key components of executive control is the ability to cancel or inhibit habitual responses. Motor response inhibition is critical in everyday life, for example, to stop crossing the street when a speeding car appears. In patients with PD, the failure of these inhibitory control mechanisms may manifest, for example, as an inability to stop festinating gait or as impulsively jumping out of a chair and losing balance. Beyond the failure of stopping or inhibiting motor responses, patients with PD are also prone to impulsivity and compulsions, leading to behaviors such as overeating or gambling. Approximately 15-20% of PD patients are diagnosed with impulse control disorders which can be exacerbated by dopaminergic medications. Furthermore, PD patients with deep brain stimulation (DBS) may develop additional impairments in executive function. Given the prevalence of executive dysfunction, the everyday-importance of this issue, and the connection with PD therapies, disease- or therapy-induced alterations in inhibitory control are an important area of research in PD.

The primary clinical objective for DBS therapy in PD has been to optimize motor function. The effect of stimulation on cognition and behavior, particularly in the subthalamic nucleus (STN), has been controversial. Behavioral side effects have been supported by reports of worsened cognition, increased impulsivity and even suicidal behavior. While large, randomized trials do not show significant detrimental changes in global cognition with DBS, meta-analyses and systematic reviews have shown adverse effects on executive functions, particularly response inhibition. Based on animal studies, the STN can be divided into a sensorimotor (dorsolateral), cognitive-associative (ventromedial) and limbic (medial) parts. Most DBS leads implanted into the STN contain four ring-shaped contacts, spaced over a total distance of 7.5-10.5mm. While surgeons generally target the dorsolateral sensorimotor region of the STN, the most ventral DBS contacts almost inevitably end up in the ventral associative or limbic regions of the nucleus. There are anecdotal observations of abrupt mood and behavioral changes (impulsivity, hypomania, depression) with STN DBS, perhaps due to spread of stimulation to the ventral STN regions. However, the effect of stimulation location on cognitive function is poorly understood and unaccounted for in clinical programming which may lead to suboptimal gains in quality of life.

Electrophysiology and imaging studies have demonstrated that the STN is a key node in the inhibitory network, although other basal ganglia nuclei are involved. The STN receives input from prefrontal cortical areas (via the prefrontal hyperdirect pathway) and is thought to provide a global inhibitory signal to the basal ganglia and thalamus to halt habitual responses and allow additional processing time in situations of conflict and uncertainty. STN DBS might (antidromically) disrupt the inhibitory signal from the cortex, leading to impulsive responses and inability to inhibit actions. However, it remains unclear whether stimulation in the STN worsens or improves motor response inhibition. It is also possible that some aspects of inhibitory control (proactive vs. reactive) can worsen during stimulation while others improve suggesting that the effects may be mediated by different pathways or mechanisms. Proactive inhibition refers to preparatory mechanisms that facilitate action inhibition (i.e. enables a person to act with restraint), while reactive inhibition is a sudden stopping process triggered by an external stimulus.

This study will address the following knowledge gaps:

1. Which cortical mechanisms (on the level of population-based electrophysiologic activity) are engaged in different aspects of inhibitory control (proactive control vs reactive; discrete movements vs continuous) in PD patients compared to healthy controls?
2. Does the effect of STN DBS on motor response inhibition depend on activation of the prefrontal hyperdirect pathway?

Successful completion of the proposed studies will provide substantial new knowledge about the frontal brain areas involved in inhibitory control, their topographic representation within the STN and means of cortico-subcortical communication. The results may inform future DBS targeting and programming strategies, aiming to avoid cognitive side effects of STN DBS. Recent engineering upgrades to clinical devices (e.g. segmented leads) allow more precise fine tuning of the stimulation field which can serve to design stimulation strategies that maximize motor benefit and minimize cognitive and behavioral side effects.

This study will enroll patients with Parkinson's Disease as well as health controls. Participation in this trial does not affect patient's clinical management. Patients' medication (levodopa) dosages and decision to undergo deep brain stimulation surgery are based on clinical needs.

There are 3 study aims:

Aim 1: To determine the effect of the PD disease process, levodopa treatment, and cognitive status on performance and cortical electrophysiology during motor response inhibition tasks. Participants with PD prior to surgery to implant the DBS leads and healthy controls are examined in Aim 1.

Aim 2: To characterize cortico-subthalamic connectivity during proactive motor response inhibition during surgery to implant clinically-indicated DBS leads in participants with PD.

Aim 3: To determine if activation of the prefrontal cortico-STN hyperdirect pathway impairs response inhibition in participants with PD from Aim 1 after implantation of DBS leads.

The experimental interventions considered in this study are: 1) medication state (PD patients are tested in levodopa-off and levodopa-on state), and 2) DBS stimulation settings (PD patients are tested under 4 stimulation settings: clinical, sham, maximizing prefrontal activation, and minimizing prefrontal activation). Healthy controls will attend two study visits, while patients with PD will be in the study for up to 18 months.

ELIGIBILITY:
Inclusion Criteria for Persons with Parkinson's Disease for Aim 1:

* diagnosis of idiopathic Parkinson's disease (PD)
* Hoehn and Yahr (H&Y) stage 2-4 (off medication)

Exclusion Criteria for Persons with Parkinson's Disease for Aim 1:

* severe tremor at rest or severe dyskinesia which would cause significant artifacts in electrophysiological signals
* inability to hold antiparkinsonian medications for research recordings
* dementia
* non-English speaker

Inclusion Criteria for Persons with Parkinson's Disease for Aim 2:

* diagnosis of idiopathic PD
* there is a clinical indication for DBS surgery
* normal preoperative MRI
* ability to tolerate microelectrode-guided neurosurgery in an awake state

Exclusion Criteria for Persons with Parkinson's Disease for Aim 2:

* presence of a coagulopathy
* uncontrolled hypertension
* heart disease
* other medical conditions considered to increase the patient's risk for surgical complications

Inclusion Criteria for Persons with Parkinson's Disease for Aim 3:

* diagnosis of idiopathic PD
* functioning DBS system

Exclusion Criteria for Persons with Parkinson's Disease for Aim 3:

* severe tremor at rest or severe dyskinesia which would cause significant artifacts in electrophysiological signals
* inability to hold antiparkinsonian medications for research recordings
* inability to tolerate temporary discontinuation of DBS therapy or alteration of stimulation settings for research purposes
* other medical conditions considered to increase the patient's risk for surgical complications

Inclusion Criteria for Healthy Controls:

* age 45-75

Exclusion Criteria for Healthy Controls:

* history of a neuropsychiatric disorder and/or treatment with psychotropic medications
* non-English speaker

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Response Time During Go/No-Go (GNG) Task for Participants in Aim 1 | Day 1 (before and after levodopa dosage for persons with PD)
  The GNG task is a tool for measuring impulsiveness by asking participants to respond to a cue signal for pressing a button. There are Go trials, where the button should be pressed, and No-Go trials, where the button should not be pressed. A total of 240 trials will be administered (5 blocks of 30) after an initial practice block (12 trials). An additional 120 Go only trials will be administered prior to the Go/No-Go blocks and serve as a control without inhibitory demands. Participants with PD attend a single study visit, completing this task twice: once after not taking PD medications for 12 hours and again after levodopa dosage. Healthy controls complete the task twice during one study visit. Response time is measured in milliseconds (ms) during the GNG task.
Percent of Errors During Go/No-Go (GNG) Task for Participants in Aim 1 | Day 1 (before and after levodopa dosage for persons with PD)
  The GNG task is a tool for measuring impulsiveness by asking participants to respond to a cue signal for pressing a button. There are Go trials, where the button should be pressed, and No-Go trials, where the button should not be pressed. A total of 240 trials will be administered (5 blocks of 30) after an initial practice block (12 trials). An additional 120 Go only trials will be administered prior to the Go/No-Go blocks and serve as a control without inhibitory demands. Participants with PD attend a single study visit, completing this task twice: once after not taking PD medications for 12 hours and again after levodopa dosage. Healthy controls complete the task twice during one study visit. Accuracy is measured as the percentage of errors during the GNG task.
Stopping Time During Modified Stop Signal (MSS) Task for Participants in Aim 1 | Day 1 (before and after levodopa dosage for persons with PD)
  For the MSS task, a fixation cross indicates the start of a trial. After a variable delay (300-700 ms) this signal is replaced by a green Go signal circle, prompting the subject to start to make circling movements with a computer mouse at approximately one rotation per second using dominant hand. After 500 ms the green circle is replaced by a visual countdown to when a red Stop signal appears (planned stop). In 50% of the trials, the Stop signal appears unexpectedly during the countdown (unplanned stop). A total of 120 trials will be administered (10 blocks of 12). Participants with PD attend a single study visit, completing this task twice: once after not taking PD medications for 12 hours and again after levodopa dosage. Healthy controls complete the task twice during one study visit. Stopping time is measured in milliseconds.
Response Time During Go/No-Go (GNG) Task for Participants in Aim 3 | Up to 12 months post-implantation of DBS leads
  The GNG task is a tool for measuring impulsiveness by asking participants to respond to a cue signal for pressing a button. There are Go trials, where the button should be pressed, and No-Go trials, where the button should not be pressed. A total of 240 trials will be administered (5 blocks of 30) after an initial practice block (12 trials). An additional 120 Go only trials will be administered prior to the Go/No-Go blocks and serve as a control without inhibitory demands. Participants with PD attend two study visits, within a 4-week period, at 6 to 12 months after implantation of the DBS leads. Participants will not take PD medications for 12 hours prior to the study visit. During each study visit chronic DBS will be turned off and two stimulation settings will be tested at each study visit so that participants all four stimulation settings over the two study visits. Response time is measured in milliseconds (ms) during the GNG task.
Percent of Errors During Go/No-Go (GNG) Task for Participants in Aim 3 | Up to 12 months post-implantation of DBS leads
  The GNG task is a tool for measuring impulsiveness by asking participants to respond to a cue signal for pressing a button. There are Go trials, where the button should be pressed, and No-Go trials, where the button should not be pressed. A total of 240 trials will be administered (5 blocks of 30) after an initial practice block (12 trials). An additional 120 Go only trials will be administered prior to the Go/No-Go blocks and serve as a control without inhibitory demands. Participants with PD attend two study visits, within a 4-week period, at 6 to 12 months after implantation of the DBS leads. Participants will not take PD medications for 12 hours prior to the study visit. During each study visit chronic DBS will be turned off and two stimulation settings will be tested at each study visit so that participants all four stimulation settings over the two study visits. Accuracy is measured as the percentage of errors during the GNG task.
Stopping Time During Modified Stop Signal (MSS) Task for Participants in Aim 3 | Up to 12 months post-implantation of DBS leads
  For the MSS task, a fixation cross indicates the start of a trial. After a variable delay (300-700 ms) this signal is replaced by a green Go signal circle, prompting the subject to start to make circling movements with a computer mouse at approximately one rotation per second using dominant hand. After 500 ms the green circle is replaced by a visual countdown to when a red Stop signal appears (planned stop). In 50% of the trials, the Stop signal appears unexpectedly during the countdown (unplanned stop). A total of 120 trials will be administered. Participants with PD attend two study visits, within a 4-week period, at 6 to 12 months after implantation of the DBS leads. Participants will not take PD medications for 12 hours prior to the study visit. During each visit chronic DBS will be turned off and two stimulation settings will be tested so that participants all four stimulation settings over the two study visits. Stopping time is measured in milliseconds.

SECONDARY OUTCOMES:
Electroencephalogram (EEG) Signals During GNG for Participants in Aim 1 | Day 1 (before and after levodopa dosage for persons with PD)
  Cortical EEG signals are acquired simultaneously during GNG task. Trigger pulses are sent from the task computer to the EEG system indicating the stimulus onsets and subject responses (button press or mouse movement). A photodiode attached to the screen will monitor the timing of stimulus presentation synchronized to EEG.
Electroencephalogram (EEG) Signals During MSS for Participants in Aim 1 | Day 1 (before and after levodopa dosage for persons with PD)
  Cortical EEG signals are acquired simultaneously during the MSS task. Trigger pulses will be sent from the task computer to the EEG system indicating the stimulus onsets and subject responses (button press or mouse movement). The mouse spatial coordinates and data from a wrist accelerometer are recorded during the MSS task. A photodiode attached to the screen will monitor the timing of stimulus presentation synchronized to EEG.
Electrocorticography (ECoG) Signals During GNG for Participants in Aim 2 | During surgical procedure to implant clinically-indicated DBS leads (approximately 15 minutes on the single day of surgery)
  ECoG signals are recorded during interoperative administration of the GNG task. The GNG task is a tool for measuring impulsiveness by asking participants to respond to a cue signal for pressing a button. There are Go trials, where the button should be pressed, and No-Go trials, where the button should not be pressed. A photodiode is affixed to the screen to synchronize the electrophysiological recordings with stimulus onsets and, like the response button readout, inputs directly into the recording system.
Electroencephalogram (EEG) Signals During GNG for Participants in Aim 3 | Up to 12 months post-implantation of DBS leads
  Cortical EEG signals are acquired simultaneously during GNG task. Trigger pulses are sent from the task computer to the EEG system indicating the stimulus onsets and subject responses (button press or mouse movement). A photodiode attached to the screen will monitor the timing of stimulus presentation synchronized to EEG.
Electroencephalogram (EEG) Signals During MSS for Participants in Aim 3 | Up to 12 months post-implantation of DBS leads
  Cortical EEG signals are acquired simultaneously during the MSS task. Trigger pulses will be sent from the task computer to the EEG system indicating the stimulus onsets and subject responses (button press or mouse movement). The mouse spatial coordinates and data from a wrist accelerometer are recorded during the MSS task. A photodiode attached to the screen will monitor the timing of stimulus presentation synchronized to EEG.

CONTACTS AND LOCATIONS:
Overall Officials: Svjetlana Miocinovic, MD, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Emory Brain Health Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported from this study will be made available for sharing with other researchers, after de-identification.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available for sharing immediately following publication and ending 5 years following article publication.
Access Criteria: Data will be available for sharing with researchers who wish to access the data, for any purpose. Requests should be directed to the corresponding author listed in the published journal article.